CLINICAL TRIAL: NCT05177341
Title: Investigating Whether Phantom Sensation Affects Autocorrelation Features of Individuals With Unilateral Below-Knee Amputation
Brief Title: Investigating The Effect of Phantom Sensation on Gait in Individuals With Unilateral Below-Knee Amputation
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Trakya University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Hilal Hotaman, PhD, Assoc Prof, Trakya University
Other Study IDs: TÜTF-BAEK 2018/451
Record Dates: First submitted 2021-12-15; First posted 2022-01-04 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2021-12

CONDITIONS: Amputation, Traumatic; Phantom Sensation
Keywords: Amputation; Phantom Sensation; Gait; Autocorrelation Function
MeSH Terms: conditions — Amputation, Traumatic; Phantom Limb

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Amputees with acceptable phantom sensation
  Interventions: Other: Determining Preferred Walking Speed
- Amputees with no phantom sensation
  Interventions: Other: Determining Preferred Walking Speed
- Control group
  Interventions: Other: Determining Preferred Walking Speed

INTERVENTIONS:
Other: Determining Preferred Walking Speed — In the beginning, sensors of the gait analysis system (RehaGait®), which can record the time-distance characteristics of consecutive multiple steps (step length, step width, double step length, and timing information, etc.) will be installed. The 7 sensors of this system are attached to the shoes of the individual, proximal to the ankle, distal thigh, and sacroiliac joint level (Aminian et al., 2014). Individuals will be required to wear casual athletic shoes and comfortable, non-knee-covering shorts. Next; Each individual will walk freely on the treadmill at their own pace. To find the preferred walking speed of the individual, Hinton et al. protocol will be used (Hinton et al., 2018). The speed of the treadmill will be increased or decreased in line with the direction of the participants. After being determined according to the protocol, the individual will practice walking at this speed for 4-5 minutes. The individual will rest as much as he or she wants.

SUMMARY:
Amputation is a problem that can be encountered for many reasons, can cause functional disability in varying severities and puts a multifaceted financial burden on individuals, society, and states. The phantom feeling is the state of the sensory sensation of a limb that does not already exist and is observed in various forms in individuals with amputation.

The aim of this project is to investigate whether the phantom sensation affects autocorrelation of gait in unilateral amputated individuals and thus to determine whether the phantom sensation is a functional sensation that affects the multifaceted nature of gait. In addition, the measurement of whether phantom sensation contributes to the ability of amputees to adapt to changing conditions and obtaining a unique calculation method that determines autocorrelation are other specific aspects of the study. The study will be conducted on individuals with unilateral traumatic transtibial amputation who have acceptable phantom sensation, individuals with no-phantom sensation and healthy individuals. Individuals who meet the inclusion criteria will be included in the gait assessment. During the evaluation, at least 512 consecutive steps will be collected from each individual when walking on the treadmill at their preferred speed. The walk test will then be repeated on the perturbation treadmill of 5-10%. It will be determined whether the gait characteristics obtained by gait analysis show autocorrelation by using signal processing methods.

DETAILED DESCRIPTION:
Amputation is a problem that can be encountered for many reasons, can cause functional disability in varying severities and puts a multifaceted financial burden on individuals, society, and states. The phantom feeling is the state of the sensory sensation of a limb that does not already exist and is observed in various forms in individuals with amputation.

The aim of this project is to investigate whether the phantom sensation affects autocorrelation of gait in unilateral amputated individuals and thus to determine whether the phantom sensation is a functional sensation that affects the multifaceted nature of gait. In addition, the measurement of whether phantom sensation contributes to the ability of amputees to adapt to changing conditions and obtaining a unique calculation method that determines autocorrelation are other specific aspects of the study. The study will be conducted on individuals with unilateral traumatic transtibial amputation who have acceptable phantom sensation, individuals with no-phantom sensation and healthy individuals. Individuals who meet the inclusion criteria will be included in the gait assessment. During the evaluation, at least 512 consecutive steps will be collected from each individual when walking on the treadmill at their preferred speed. The walk test will then be repeated on the perturbation treadmill of 5-10%. It will be determined whether the gait characteristics obtained by gait analysis show autocorrelation by using signal processing methods.

ELIGIBILITY:
Group 1 (amputated individuals with phantom sensation) inclusion criteria:

* Having an acceptable (non-irritating) phantom sensation that persists throughout the day, even if the severity is variable
* Having unilateral below-knee amputation due to trauma
* Using OttoBock® prosthesis with dynamic foot component, silicone liner design and active vacuum system: The reason for choosing this prosthesis; This is because it is a prosthesis documented in the literature, with the highest standards of use in today's conditions, the most preferred in the international platform, used in research, and advantageous for use in daily life. Thus, deficiencies that may arise from the design of the prosthesis will not be encountered.
* At least 2 years have passed since amputation surgery
* Using the last prosthesis for at least 6 months for at least 6-8 hours a day
* Being within the limits of body mass index (weight/height2: 18.5-24.9 kg/m2) accepted as normal by the World Health Organization
* Having the ability to speak and understand Turkish
* Not having any balance and coordination difficulties that can be observed with clinical functional tests
* Not having any joint contracture or muscle shortness that may affect walking ability
* Agree to participate in the study

Group 1 (amputated individuals with phantom sensation) exclusion criteria:

* Undergoing amputation surgery for non-traumatic reasons
* Having multiple amputations
* To be followed up with any medical pre-diagnosis (orthopedic, neurological, cardiovascular, psychiatric, etc.)
* To be followed up with any medical diagnosis (orthopedic, neurological, cardiovascular, psychiatric, etc.)
* Being on medication during the research
* Having consumed alcohol in the last 48 hours
* Taking painkillers in the last 48 hours
* Having a history of surgery and acute trauma in the last 6 months
* Having a history of falling in the last 1 year
* Loss of sensation in the remaining limb (stump) after amputation
* Having a disturbing phantom feeling
* Having any chronic and/or acute pain, including phantom pain and stump pain
* Observing any shortness, contracture or balance problems in the pre-tests

Group 2 - (amputated individuals without phantom sensation) inclusion criteria:

* Having unilateral below-knee amputation due to trauma
* Volunteering to participate in the study
* Using OttoBock® prosthesis with dynamic foot component, silicone liner design and active vacuum system (Picture 1)
* At least 2 years have passed since amputation surgery
* Using the last prosthesis for at least 6 months for at least 6-8 hours a day
* Being within the limits of body mass index (weight/height2: 18.5-24.9 kg/m2) accepted as normal by the World Health Organization
* Having the ability to speak and understand Turkish
* Absence of phantom sensation at any time and movement in the last 4 weeks

Group 2 - (amputated individuals without phantom sensation) exclusion criteria:

* Undergoing amputation surgery for non-traumatic reasons
* Having multiple amputations
* To be followed up with any medical pre-diagnosis (orthopedic, neurological, cardiovascular, psychiatric, etc.)
* To be followed up with any medical diagnosis (orthopedic, neurological, cardiovascular, psychiatric, etc.)
* Being on medication during the research
* Having consumed alcohol in the last 48 hours
* Taking painkillers in the last 48 hours
* Having a history of surgery and acute trauma in the last 6 months
* Having a history of falling in the last 1 year
* Loss of sensation in the remaining limb (stump) after amputation
* Having a phantom feeling
* Having any chronic and/or acute pain, including phantom pain and stump pain
* Observing any shortness, contracture or balance problems in the pre-tests

Group 3 - (healthy volunteers) inclusion criteria:

* Being within the limits of body mass index (weight/height2: 18.5-24.9 kg/m2) accepted as normal by the World Health Organization
* Having the ability to speak and understand Turkish
* Agree to participate in the study

Group 3 - (healthy volunteers) exclusion criteria:

* To be followed up with any medical pre-diagnosis (orthopedic, neurological, cardiovascular, psychiatric, etc.)
* To be followed up with any medical diagnosis (orthopedic, neurological, cardiovascular, psychiatric, etc.)
* Being on medication during the research
* Having consumed alcohol in the last 48 hours
* Taking painkillers in the last 48 hours
* Having a history of surgery and acute trauma in the last 6 months
* Having a history of falling in the last 1 year
* Observing any shortness, contracture or balance problems in the pre-tests

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Traumatic transtibial amputees or age and gender matched healthy individuals
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-01 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Gait Analysis on Flat Ground | 5 minutes after the protocol for determining the preferred walking speed
  In order to collect the data required for the autocorrelation calculation in flat walking, the subject will be placed on the treadmill (REAX RUN) and he or she will be asked to continue his walking at the "preferred speed" level obtained with the previous protocol, until at least 512 steps are collected. This walk is expected to take 3-4 minutes in total. After a sufficient number of steps is reached, the treadmill will be gradually slowed down and stopped. Afterward, the individual will be taken to rest again.
Gait analysis on Perturbed Ground | 5 minutes after walking on the flat ground
  After the resting period is terminated, the individual will start walking at the speed determined according to the Hinton protocol on the treadmill (REAX RUN) for gait analysis again. During the second walk, 5-10% perturbation will be given on the treadmill until 512 steps are collected. The autocorrelation analysis to be performed with the data taken during walking on the perturbed ground will measure the adaptability of the individual's gait to changing conditions. The data of the walk will be automatically saved on the system computer. Whether the autocorrelation feature of the gait is observed or not will be calculated mathematically using signal processing methods.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hinton DC, Cheng YY, Paquette C. Everyday multitasking habits: University students seamlessly text and walk on a split-belt treadmill. Gait Posture. 2018 Jan;59:168-173. doi: 10.1016/j.gaitpost.2017.10.011. Epub 2017 Oct 7. PMID 29032000
- [Background] Aminian K, Dadashi F, Mariani B, Lenoble-Hoskovec C, Santos-Eggimann B, Büla CJ. Gait analysis using shoe-worn inertial sensors: how is foot clearance related to walking speed? Proceedings of the 2014 ACM international joint conference on Pervasive and ubiquitous computing. 2014; 481-485.